CLINICAL TRIAL: NCT07085923
Title: Dietary Counselling And Exercise To Combat Cardiovascular Disease Risk In Norwegian Patients With A Severe Mental Illness
Brief Title: Norwegian Mental Illness Heart Health Study
Acronym: NORMI-Heart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Madeleine Elisabeth Angelsen (Other)
Responsible Party: Sponsor-Investigator, Madeleine Elisabeth Angelsen, PhD Fellow under the supervision of Professor Kjetil Retterstøl, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108677
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-07

CONDITIONS: Cardio Vascular Disease; Metabolic Syndrome (MetS); Severe Mental Disorder; Schizophrenia and Schizophrenia Spectrum Psychosis; Bipolar Disease Type I; Overweight and/or Obesity; CVD Risk Factors; Severe Mental Illness
Keywords: Severe Mental Illness; Cardiovascular Disease; Lifestyle Intervention; Healthy Diet; Exercise; CVD-risk; Schizophrenia; Antipsychotic Medication; Bipolar Disorder; Non-pharmacological intervention; Clinical Dietitian
MeSH Terms: conditions — Metabolic Syndrome; Mental Disorders; Schizophrenia; Cardiovascular Diseases; Motor Activity; Bipolar Disorder | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel assignment of participants to intervention or control group in a 1:1 ratio, stratified by diagnosis. The initial control group is offered the intervention after 6 months, without outcome assessments, for ethical reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): Participants in this arm receive a 6-month lifestyle program in addition to usual mental health care. The intervention includes monthly individual sessions with a clinical dietitian, omega-3 supplementation, monthly group-based physical activity sessions led by an instructor, and support to follow a personalized training plan.
  Interventions: Behavioral: Lifestyle Intervention
- Control (No Intervention): Participants in this arm receive treatment as usual (TAU) in mental health care. After the 6-month study period, they are offered the same lifestyle program without data collection, for ethical reasons.

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The Lifestyle Program consists of monthly one-on-one dietary counselling sessions with a registered clinical dietitian, monthly group-based physical activity sessions led by an instructor, and support to follow a personalized exercise plan. The intervention focuses on cardioprotective dietary changes, weight reduction, and increasing physical activity at moderate-to-high intensity to meet recommended amount. Participants will receive dietary supplementation corresponding to a therapeutic dose of 1000 mg EPA+DHA per day from fish oil. During monthly visits with the dietitian, data will be collected to monitor progress and support adherence. Participants will be encouraged to monitor body weight at home between visits (bathroom scales are loaned as needed), and follow up is carried out biweekly via phone-calls. The intervention is designed to be feasible within routine mental health care and tailored to the needs of adults with severe mental illness.
  Other Names: Dietary Counselling and Exercise; Lifestyle Program
  Arms: Lifestyle Intervention

SUMMARY:
Norwegian patients with severe mental illnesses (SMI), such as schizophrenia spectrum or bipolar disorder, lose on average 10 years of life compared to mentally healthy individuals. Much of this gap is due to heart disease. Unhealthy lifestyle habits, including poor diet and physical inactivity, contribute to higher levels of metabolic risk factors for heart disease in this population.

The goal of this clinical trial is to find out if a lifestyle program including dietary counselling and regular physical exercise can help people with SMI to improve their physical and mental health.

The main questions it aims to answer are:

* Does adherence to a healthy lifestyle program lead to reduced estimated risk of heart disease?
* Does it change lifestyle habits, body weight and composition, and metabolic risk markers over six months?
* Can participants with severe mental illness complete a healthy lifestyle program, and do they find it acceptable?

Researchers will compare two groups: one that receives the lifestyle program in addition to regular mental health care, and one that receives regular care only.

During the six month program, participants in the lifestyle group will:

* Meet with a clinical dietitian once a month for dietary counselling
* Take part in group-based physical activity sessions once a month, and receive support to follow a personal training plan

Around 70 adults will take part in the study. The results may help improve the way lifestyle support is offered to people living with severe mental illness and inform health care providers about strategies to improve physical health in this vulnerable group.

DETAILED DESCRIPTION:
People with severe mental illness (SMI) such as schizophrenia spectrum- or bipolar disorder face a markedly increased risk of early death compared to the general population, with cardiovascular disease (CVD) as the leading cause. This excess risk is partly explained by modifiable lifestyle-related risk factors such as physical inactivity, poor diet quality, and the metabolic side effects of antipsychotic medication. Despite this, people with SMI often receive less preventive somatic care and limited support to adopt healthier habits.

The scientific evidence for the effectiveness of lifestyle interventions in this population is still limited, and previous trials have yielded mixed results. The most promising studies have combined professional dietary counselling with physical activity at moderate to high intensity. This study builds on previous research and clinical experience with the patient group, and responds to a documented need for targeted, feasible interventions in mental health services.

The study aims to contribute to the evidence base by testing a feasible, multidisciplinary intervention integrated in routine mental health care. This randomized controlled trial (RCT) will evaluate the impact of a structured lifestyle program on the estimated CVD risk and associated metabolic and lifestyle outcomes in Norwegian adults with an SMI.

Participants will be randomized in a 1:1 ratio to either a 6-month lifestyle intervention or a control group receiving treatment as usual (TAU) in mental health care. The study will include approximately 70 overweight adults with schizophrenia spectrum (ICD-10 F20-29) or bipolar disorder (ICD-10 F31). For ethical reasons, the control group will be offered the same lifestyle program after the 6-month trial period, without accompanying data collection.

The intervention period lasts six months and consists of:

* Monthly one-on-one sessions with a registered clinical dietitian, focused on cardioprotective dietary changes, practical food strategies, and weight reduction.
* Monthly group-based physical activity sessions led by an instructor, tailored to the participants' physical capacity.
* Support to follow a personalized training plan meeting the recommended amount of physical activity on moderate-high intensity.

The intervention is designed to integrate into existing mental health services and accommodate the needs and challenges specific to people with SMI, such as medication side effects, low energy levels, and cognitive symptoms. User panels including patients with lived experiences are involved in tailoring the intervention. Fidelity and feasibility will be evaluated through structured feedback and attendance records.

The study will assess whether adherence to a healthy lifestyle, measured with the DIGIKOST Lifestyle Index, affects estimated 10-year CVD risk, using a validated risk prediction tool. Weight monitoring, blood pressure recordings and blood test results are incorporated in the risk prediction, and this data will be assessed regularly throughout the study period. Secondary outcomes include changes in objectively measured physical activity (accelerometer), adherence to national lifestyle recommendations and diet quality (measured with a validated food frequency questionnaire, DIGIKOST), body composition (Bioelectrical impedance), waist circumference, body weight, and relevant biomarkers including blood lipids and glucose, in the intervention group compared to TAU. The presence of metabolic syndrome will also be evaluated using IDF and ATP III criteria. Health-related quality of life will be measured using a simple and validated questionnaire (PROMIS-29).

Statistical analysis will follow the intention-to-treat principle and use linear mixed-effects models to evaluate between-group changes from baseline to 6 months. In addition, interim measurements at 3 months will be used for secondary analyses to assess early changes, explore the trajectory of intervention effects, and monitor adherence and retention. This mid-intervention timepoint is also collected in the control group to enable temporal comparisons and better understand the dynamics of lifestyle change in both groups. Exploratory analyses will investigate predictors of adherence, effect heterogeneity, and timing of response.

The trial is part of a PhD project and will contribute to improved understanding of how lifestyle interventions can be tailored and implemented to improve physical health in people with SMI. The findings may help inform future clinical practice and reduce somatic health disparities in this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of F20-29 (schizophrenia spectrum) or F31 (bipolar affective disorder)
* Current use of antipsychotic medication (first- or second generation) or lithium
* Body Mass Index > or = 27 kg/m^2

Exclusion Criteria:

Psychiatric condition:

* Inability to provide informed consent*
* Acute psychiatric crisis*
* Significant cognitive impairment* *These criteria will be evaluated and confirmed by the participant's primary mental health care provider before enrollment

Medication initiated during the intervention period:

* GLP-1 receptor agonists
* Antihypertensive medication
* Antidiabetic medication
* Lipid-lowering medication

Alcohol consumption:

-More than 14 units per week (men) or more than 7 units per week (women)

Somatic conditions:

* Type 1 diabetes
* Established cardiovascular disease
* Body Mass Index (BMI) <27 kg/m²
* Pregnancy
* Inability to perform physical exercise

Somatic risk findings at baseline:

* HbA1c >57 mmol/mol (7.4%)
* LDL cholesterol >5.0 mmol/L
* Blood pressure >180/100 mmHg
* Active malignant disease

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Estimated Risk of Heart Disease (QRISK3) | From baseline to 6 months
  Compare the change in estimated cardiovascular disease risk between intervention and control (Treatment as Usual) groups over 6 months, using the validated QRISK3 algorithm.
Association Between Change in Lifestyle Adherence and Change in QRISK3 Score | From baseline to 6 months
  Explore whether change in adherence to a healthy lifestyle, measured with the DIGIKOST Lifestyle Index, predicts change in estimated cardiovascular disease risk (QRISK3).

SECONDARY OUTCOMES:
Change in Objectively Measured Physical Activity (Accelerometer) | From baseline to 6 months
  Physical activity will be assessed using a thigh-worn accelerometer worn for 7 consecutive days at baseline and again after 6 months. The device captures activity intensity and duration, including time spent sedentary, standing, and in moderate-to-vigorous physical activity. Between-group differences will be analyzed to evaluate the impact of the lifestyle intervention.
Change in lifestyle adherence score (DIGIKOST Lifestyle Index) | Baseline and 6 months
  Healthy lifestyle adherence will be measured using the DIGIKOST Lifestyle Index at baseline and 6 months. The index serves as a proxy for behavioral change. Between-group differences (intervention vs. control) in change from baseline will be evaluated after the intervention (6 months)
Change in Diet Quality (DIGIKOST Diet Index and 24-Hour Dietary Recall) | From baseline to 6 months
  Assess changes in diet quality based on a validated food frequency questionnaire (DIGIKOST Diet Index) and nutritional composition measured with 24-hour dietary recalls (repeated by phone call for validity), relative to Norwegian dietary recommendations. Repeated at baseline and after 6 months
Presence and Change in Metabolic Syndrome (IDF and ATP-III Criteria) | Baseline, 3 months and 6 months
  Metabolic syndrome will be assessed at baseline, 3 months, and 6 months using both the International Diabetes Federation (IDF) and the Adult Treatment Panel III (ATP-III) diagnostic criteria. Between-group differences (intervention vs. control) in the prevalence and change in metabolic syndrome status from baseline will be evaluated at 3 and 6 months.
Change in Blood Biomarkers Related to Cardiometabolic Health | From baseline, at 3 months and after 6 months
  Fasting blood samples will be collected at baseline, 3 months, and 6 months to evaluate changes in cardiometabolic and nutritional biomarkers. Participants will be instructed to fast for at least 8 hours and avoid alcohol and vigorous physical activity for 24 hours prior to sampling. Samples will be drawn by the PhD candidate. Biomarkers include total cholesterol, LDL, HDL, triglycerides, ApoB, Lp(a), glucose, HbA1c, ALAT, ferritin, folate, vitamin D, homocysteine, hs-CRP, hydroxybutyrate, and acetoacetate. Between-group differences (intervention vs. control) in changes from baseline will be assessed at 3 and 6 months. The 3-month time point enables evaluation of early physiological responses to the intervention. Data will also be used to determine the presence and change in metabolic syndrome based on standard criteria.
Change in Body Weight | Baseline, 3 months, and 6 months
  Body weight will be measured at baseline, 3 months, and 6 months in both groups to assess between-group changes (intervention vs. treatment as usual). In the intervention group, additional monthly measurements will be conducted to track individual progress throughout the intervention period. A calibrated digital scale validated for clinical and research use will be used. Participants will be instructed to wear light clothing, remove shoes, and avoid eating or drinking for at least 8 hours prior to measurement.
Change in Waist Circumference | Baseline, 3 months and 6 months
  Waist circumference will be measured with a measuring tape at the midpoint between the lowest rib and the iliac crest. Measurements will be conducted at baseline, 3 months, and 6 months in both groups to assess between-group differences (intervention vs. treatment as usual). In the intervention group, additional monthly measurements will be performed to monitor changes over time.
Change in Blood Pressure | Baseline, 3 months, and 6 months
  Systolic and diastolic blood pressure will be measured in a seated position using automated equipment. Measurements will be taken at baseline, 3 months, and 6 months in both groups to evaluate between-group changes (intervention vs. treatment as usual). In the intervention group, additional monthly measurements will be conducted to track individual progress throughout the intervention period.
Change in Body Composition (BIA) | Baseline, 3 months and 6 months
  Body composition will be assessed using a bioelectrical impedance analysis (BIA) device validated for research purposes, at baseline, 3 months, and 6 months in both groups to evaluate changes in fat mass, fat-free mass, and total body weight. In the intervention group, BIA will also be performed monthly to track individual changes throughout the intervention period.

OTHER OUTCOMES:
Change in Health-Related Quality of Life (PROMIS-29) | Baseline, 3- and 6 months
  Assess changes in self-reported health-related quality of life using the PROMIS-29 instrument, a validated questionnaire covering physical, mental, and social functioning, in the intervention group compared to treatment as usual. Between-group differences in change from baseline will be evaluated at 3- and 6 months.
Feasibility and Acceptability of the Lifestyle Program (qualitative) | Throughout the 6 month intervention period
  Explore participants' experiences and the perceived feasibility and acceptability of the lifestyle intervention. Data will be collected through field notes, informal participant feedback, and illustrative quotes during dietitian consultations and group sessions. Notes will be recorded continuously by the clinical dietitian and physical activity instructor throughout the 6-month intervention period.
Predictors of adherence and effect heterogeneity | Baseline to 6 months
  Exploratory analyses will investigate whether baseline characteristics such as diagnosis, sex, BMI, and type of medication predict adherence or modify the effect of the intervention. Analyses will also assess differential responses within subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Kjetil Retterstøl, Professor, MD, Principal Investigator — University of Oslo
Locations (1):
- Department for nutrition science, Domus Medica, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rocks T, Teasdale SB, Fehily C, Young C, Howland G, Kelly B, Dawson S, Jacka F, Dunbar JA, O'Neil A. Effectiveness of nutrition and dietary interventions for people with serious mental illness: systematic review and meta-analysis. Med J Aust. 2022 Oct 2;217 Suppl 7(Suppl 7):S7-S21. doi: 10.5694/mja2.51680. PMID 36183316
- [Background] Gurusamy J, Gandhi S, Damodharan D, Ganesan V, Palaniappan M. Exercise, diet and educational interventions for metabolic syndrome in persons with schizophrenia: A systematic review. Asian J Psychiatr. 2018 Aug;36:73-85. doi: 10.1016/j.ajp.2018.06.018. Epub 2018 Jun 30. PMID 29990631
- See also: This page from the Norwegian Directorate of Health presents the recommended national care pathway for adults with mental illness, including guidance on somatic screening and treatment to ensure coordinated, high-quality, and equitable health services. — https://www.helsedirektoratet.no/nasjonale-forlop/psykiske-lidelser-voksne/bakgrunn-metode-og-prosess

DOCUMENTS (1):
  • Informed Consent Form (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT07085923/ICF_000.pdf